CLINICAL TRIAL: NCT07077174
Title: Effects of PERMISSive Lung-protective Ventilation on Outcome in Critically Ill Invasively Ventilated Patients (PERMISS) - a Feasibility and Safety Pilot Study for a Randomized Clinical Trial
Brief Title: Effects of PERMISSive Lung-protective Ventilation on Outcome in Critically Ill Invasively Ventilated Patients
Acronym: PERMISS pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier de Graaf Groep (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-009624.P25.028; NL-OMON57603 (Other: Overzicht van Medisch-wetenschappelijk Onderzoek in Nederland (OMON))
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation; Acute Hypoxemic Respiratory Failure; Intensive Care (ICU)
Keywords: mechanical ventilation; intensive care unit; mechanical power; respiratory rate
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Permissive lung-protective ventilation (Experimental): The goal is to achieve the lowest possible respiratory rate (RR) according to a guideline < 1 hour after start of ventilation in the ICU.
  Interventions: Other: Permissive lung-protective ventilation
- Conventional lung-protective ventilation (Active Comparator): The respiratory rate is set according to standard of care < 1 hour after start of ventilation in the ICU.
  Interventions: Other: Conventional lung-protective ventilation

INTERVENTIONS:
Other: Permissive lung-protective ventilation — The goal is to achieve the lowest possible respiratory rate (RR) according to a guideline in which the target RR is estimated by combining the baseline RR with the results of arterial blood gas analysis (ABG), determined by the highest acceptable partial pressure of carbon dioxide (PaCO2) of ≤ 8.5 kPa (64 mmHg) but limited by the lowest acceptable arterial pH (pHa) of > 7.20. The RR is gradually decreased, in steps of 2 breaths every 10 minutes, based on continuous end-tidal CO2 monitoring. To ensure that the pHa does not fall below 7.20, following randomization, ABGs are repeated every hour until the target RR is reached, for at least 6 hours. Thereafter, blood gas analyses are repeated at least every 8 hours (at the start of every nursing shift). Down-titration of RR stops at a rate of 4 breaths per minute. This approach continues until the switch to spontaneous breathing. Of note, when the pHa is > 7.50, this must first be decreased to ≤ 7.50 based on local protocol.
  Arms: Permissive lung-protective ventilation
Other: Conventional lung-protective ventilation — Following randomization, which should happen within 1 hour after start of ventilation in the ICU, the RR is set according to standard of care, based on continuous end-tidal CO2 monitoring, to target a normal PaCO2 (4.7-6.4 kPa or 35-48 mmHg) combined with a pHa within the range of 7.35 to 7.45. Following randomization, blood gas analyses are repeated every hour for at least 6 hours, and thereafter at least every 8 hours (at the start of every nursing shift). This approach continues until the weaning phase.
  Arms: Conventional lung-protective ventilation

SUMMARY:
RATIONALE Lung-protective ventilation using a lower respiratory rate (RR) is an appealing strategy to reduce ventilation intensity, which may require permissive hypercapnia. However, the feasibility and safety of this so-called 'permissive lung-protective ventilation' must be investigated, before conducting a large randomized clinical trial to evaluate its effectiveness on patient-centered outcomes.

OBJECTIVE To study the feasibility and safety of permissive lung-protective ventilation in adult critically ill patients receiving invasive ventilation for acute hypoxemic respiratory failure, and to inform the design of a future randomized clinical trial in this patient population.

HYPOTHESIS Permissive lung-protective ventilation is a feasible and safe ventilation strategy.

STUDY DESIGN Multicenter, randomized clinical pilot trial. STUDY POPULATION Critically ill patients, aged > 18 years, intubated for acute hypoxemic respiratory failure, and expected to receive ventilation for > 24 hours.

METHODS Patients are randomized to permissive lung-protective ventilation wherein RR is stepwise reduced, or to conventional lung-protective ventilation.

OUTCOME MEASURES The primary endpoint is feasibility, assessed by the difference in respiratory rate (RR) between the two groups, from the start of mechanical ventilation until first extubation. Secondary endpoints include protocol compliance and feasibility of collecting data, and safety, assessed by the occurrence of unacceptable hypercapnia and hypoxemia and the incidence of ventilator-associated complications SAMPLE SIZE To estimate the appropriate sample size for this pilot study, we considered the primary feasibility endpoint of detecting a difference in the respiratory rate (RR). Assuming an expected mean difference in RR of 7.5, based on previous studies [1, 2], with an SD of 10, a power of 90% and an alpha of 0.05, with a drop-out rate estimated at 10%, a two-tailed t-test was used. The required sample size is 84 patients (42 patients per group).

NATURE AND EXTENT OF THE BURDEN AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS Ventilation with a lower RR may require permissive hypercapnia, which, when kept within safe limits, is safe. In current daily practice, there is no guidance in setting RR; consequently, RR varies widely across patients and is often set high. This pilot study compares two forms of lung-protective ventilation, both considered standard care in current ICU practice. The control group receives conventional ventilation with low tidal volumes and high RR to maintain normal PaCO₂ and pH. The intervention group, permissive ventilation, uses a lower RR to reduce mechanical power, accepting mild hypercapnia and acidosis. Permissive ventilation is most often reserved for patients with severe lung conditions, where ventilator settings are more complex and ventilation intensity is high. In these patients, permissive ventilation is considered safe, and may even be beneficial. We aim to evaluate this strategy more broadly in critically ill patients. The collection of demographic, ventilation and outcome data causes no harm to patients. Blood is drawn for arterial blood gas analysis, but this is also part of standard care.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the participating ICUs;
* intubated and receiving invasive ventilation for acute hypoxemic respiratory failure;
* expected duration of ventilation of at least 24 hours and
* receiving invasive ventilation ≤ 1 hour.

Exclusion Criteria:

* age below 18 years;
* intubated and receiving invasive ventilation for other reasons than acute hypoxemic respiratory failure;
* receiving or planned to receive veno-venous, veno-arterial or arterio-venous extracorporeal membrane oxygenation (ECMO);
* having COPD GOLD III and IV;
* contra-indication for hypercapnia, such as ongoing cardiac ischemia (as defined in the guideline of the European Society of Cardiology), or having suspected or confirmed increased intracranial pressure due to brain injury, judged by the attending physician;
* having metabolic acidosis, with a pH < 7.20 and judged by the attending physician to have a metabolic cause;
* after cardiac resuscitation;
* any neurologic diagnosis that can prolong duration of mechanical ventilation, e.g., Guillain-Barré syndrome, high spinal cord lesion or amyotrophic lateral sclerosis, multiple sclerosis, or myasthenia gravis;
* suspected or confirmed pregnancy;
* participation in another interventional trial using similar endpoints;
* previously randomized in this study;
* no informed consent; or
* admitted for terminal care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | from the start of mechanical ventilation until first extubation, up to 28 days
  Assessed by the difference in respiratory rate (RR) between the two groups

SECONDARY OUTCOMES:
Safety of the intervention | From the start of mechanical ventilation until first extubation, up to 28 days.
  Assessed by the occurrence of unacceptable hypercapnia and hypoxemia and the incidence of ventilator-associated complications
Compliance of the protocol | From the start of mechanical ventilation until first extubation, up to 28 days.
  Determined by reflecting whether the target RR was reached and maintained during the ventilation period in the permissive lung-protective ventilation group.
Compliance of the protocol | from start of ventilation until first extubation, up to 28 days.
  Determined by how often a patient was switched back to the other ventilation group
Feasibility of collecting data | from start of mechanical ventilation until follow-up at day 90.
  assessed by the amount of missing data

CONTACTS AND LOCATIONS:
Overall Officials: Laura Buiteman-Kruizinga, RN, PhD, Principal Investigator — Reinier de Graaf Groep; Marcus J. Schultz, MD, PhD, Study Chair — Amsterdam UMC
Locations (4):
- Netherlands (3):
  - ZiekenhuisGroep Twente, Almelo
  - Reinier de Graaf Hospital, Delft
  - Dijklander Hospital, Hoorn
- Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF